CLINICAL TRIAL: NCT02436577
Title: An Open-label, Randomized, Three-period, Three-treatment, Crossover, Single-centre, Single-dose Study to Assess the Bioequivalence Between Ticagrelor Orodispersible Tablets and Ticagrelor Immediate-release Tablets in Healthy Japanese Subjects.
Brief Title: Study to Assess the Bioequivalence Between Ticagrelor Orodispersible Tablets and Ticagrelor Immediate-release Tablets in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5139C00004
Record Dates: First submitted 2015-04-07; First posted 2015-05-07 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Bioequivalence; Healthy Japanese Subjects; Pharmacokinetics
Keywords: ticagrelor orodispersible tablet; ticagrelor immediate-release tablet; bioequivalence; Phase I; healthy Japanese subjects
MeSH Terms: interventions — Water; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence ABC (Experimental): Treatment A in Period 1, Treatment B in Period 2 and Treatment C in Period 3
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 150 mL of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor IR tablet (90 mg) administered with 150 mL of water
- Sequence BCA (Experimental): Treatment B in Period 1, Treatment C in Period 2 and Treatment A in Period 3
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 150 mL of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor IR tablet (90 mg) administered with 150 mL of water
- Sequence CAB (Experimental): Treatment C in Period 1, Treatment A in Period 2 and Treatment B in Period 3
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 150 mL of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor IR tablet (90 mg) administered with 150 mL of water
- Sequence ACB (Experimental): Treatment A in Period 1, Treatment C in Period 2 and Treatment B in Period 3
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 150 mL of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor IR tablet (90 mg) administered with 150 mL of water
- Sequence BAC (Experimental): Treatment B in Period 1, Treatment A in Period 2 and Treatment C in Period 3
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 150 mL of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor IR tablet (90 mg) administered with 150 mL of water
- Sequence CBA (Experimental): Treatment C in Period 1, Treatment B in Period 2 and Treatment A in Period 3
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 150 mL of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor IR tablet (90 mg) administered with 150 mL of water

INTERVENTIONS:
Drug: Ticagrelor OD tablet (90 mg single dose) administered with 150 mL of water — Ticagrelor 90 mg OD tablet, single dose
  Other Names: Treatment A
Drug: Ticagrelor OD tablet (90 mg single dose) administered without water — Ticagrelor 90 mg OD tablet, single dose
  Other Names: Treatment B
Drug: Ticagrelor IR tablet (90 mg) administered with 150 mL of water — Ticagrelor 90 mg IR tablet, single dose
  Other Names: Treatment C

SUMMARY:
This study will be an open-label, randomised, three-period, three-treatment, crossover study in healthy Japanese male and female of non-childbearing potential subjects, performed at a single study centre.

The objective of the study is to assess the bioequivalence of ticagrelor orodispersible (OD) tablets when administered with water and without water and ticagrelor immediate-release (IR) tablets.

DETAILED DESCRIPTION:
Study to evaluate the bioequivalence of ticagrelor orodispersible (OD) tablets administered with water and without water and ticagrelor immediate-release (IR) tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 20 to 45 years with suitable veins for cannulation or repeated venepuncture.
* Be Japanese. Japanese is defined as having both parents and four grandparents who are Japanese. This includes second and third generation Japanese whose parents or grandparents are living in a country other than Japan.
* Females must have a negative pregnancy test at screening and on each admission to the clinical unit, must not be lactating, and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  * Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Have a body mass index (BMI) between 18.0 and 27.0 kg/m2 inclusive and weigh at least 45 kg and no more than 85 kg inclusive.
* Be able and willing to communicate with the investigator and comply with all study procedures, including reproductive restrictions.

Exclusion Criteria: - History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influences the results or the potential subject's ability to participate in the study.

* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* History of hemophilia, von Willebrand's disease, lupus anticoagulant, or other diseases/syndromes that can either alter or increase the propensity for bleeding.
* A personal history of vascular abnormalities including aneurysms; a personal history of severe hemorrhage, hematemesis, melena, hemoptysis, severe epistaxis, severe thrombocytopenia, intracranial hemorrhage; or rectal bleeding within 1 year prior to screening; or history suggestive of peptic ulcer disease; or at the discretion of the investigator.
* History of a clinically significant non-traumatic bleed or clinically significant bleeding risk, as judged by the investigator.
* Use of aspirin, ibuprofen, non-steroidal anti-inflammatory drugs (NSAIDs), or any other drug known to increase the propensity for bleeding for 2 weeks before randomization.
* Platelet count less than 150 x 10^9/L.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, Dr., Principal Investigator — PAREXEL Early Phase Clinical Unit London
Locations (1):
- Research Site, Harrow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL International, Early Phase Clinical Unit London, Middlesex, United Kingdom.
Pre-assignment Details: Participants were randomized to a 6 sequence Williams square design for 3 periods and 3 treatments: 90 mg ticagrelor orodispersible (OD) tablet with water (Treatment A); 90 mg ticagrelor OD tablet without water (Treatment B); 90 mg ticagrelor immediate-release (IR) tablet with water (Treatment C).
Groups:
- ABC Sequence: Subjects were administered a single dose of Treatment A, B and C as first, second and third interventions (3 days each) respectively where each intervention is separated by the washout period of minimum 7 days.
- BCA Sequence: Subjects were administered a single dose of Treatment B, C and A as first, second and third interventions (3 days each) respectively where each intervention is separated by the washout period of minimum 7 days.
- CAB Sequence: Subjects were administered a single dose of Treatment C, A and B as first, second and third interventions (3 days each) respectively where each intervention is separated by the washout period of minimum 7 days.
- ACB Sequence: Subjects were administered a single dose of Treatment A, C and B as first, second and third interventions (3 days each) respectively where each intervention is separated by the washout period of minimum 7 days.
- BAC Sequence: Subjects were administered a single dose of Treatment B, A and C as first, second and third interventions (3 days each) respectively where each intervention is separated by the washout period of minimum 7 days.
- CBA Sequence: Subjects were administered a single dose of Treatment C, B and A as first, second and third interventions (3 days each) respectively where each intervention is separated by the washout period of minimum 7 days.
Period: Overall Study
Arm/Group | ABC Sequence | BCA Sequence | CAB Sequence | ACB Sequence | BAC Sequence | CBA Sequence
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 6 | 7 | 7 | 7 | 7
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per the Participant Screening Log a total of 51 subjects underwent screening visits and 7 subjects were considered screen failures. Of the 44 subjects who were determined eligible, 1 withdrew consent and 1 was not needed as the study was filled. Hence, only 42 subjects were randomized and received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABC Sequence | BCA Sequence | CAB Sequence | ACB Sequence | BAC Sequence | CBA Sequence | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 32 (3) | 32 (9) | 32 (8) | 31 (7) | 29 (8) | 31 (7)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 7 | 7 | 7 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: Comparison of Cmax (maximum observed plasma concentration) of ticagrelor and its active metabolite AR-C124910XX following single doses of the orodispersible (OD) tablet - when administered with and without water - and ticagrelor immediate-release (IR) tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: The pharmacokinetic (PK) analysis set consisted of all participants for whom at least 1 of the primary PK parameters, for a given analyte, was calculated for at least 2 treatment periods (where 1 of the treatment periods was the period in which the participant received the reference product [Treatment C]) and who had no major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: Participants received Ticagrelor OD tablets administered with water. The OD tablet was placed with dry hands on the tongue for disintegration and was swallowed subsequently with 150 mL non-carbonated water at room temperature.
- Treatment B: Participants received Ticagrelor OD tablets administered without water. The OD tablet was placed with dry hands on the tongue for disintegration and was swallowed subsequently with saliva.
- Treatment C: Participants received Ticagrelor IR tablets administered orally with 150 mL of water.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
ng/mL
  Ticagrelor | 529 (38.4) | 534 (29.8) | 569 (37.0)
  AR-C124910XX | 165 (31.4) | 158 (36.5) | 170 (35.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Statistical Assessment of Bioequivalence for Ticagrelor Following Ticagrelor OD Tablets Compared to Ticagrelor IR Tablets; Test type: Superiority or Other; ANOVA; Geometric Mean Ratio = 93.16, 90% CI 2-sided [85.80 to 101.15]
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 93.67, 90% CI 2-sided [87.88 to 99.84]
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Statistical Assessment of Bioequivalence for metabolite AR-C124910XX Following Ticagrelor OD Tablets Compared to Ticagrelor IR Tablets; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 96.79, 90% CI 2-sided [88.27 to 106.14]
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 92.32, 90% CI 2-sided [85.04 to 100.23]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Analyte Concentration AUC (0-t) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: Comparison of AUC(0-t) (Area under the plasma concentration-time curve from time zero to time of last quantifiable analyte concentration) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: The PK analysis set consisted of all participants for whom at least 1 of the primary PK parameters, for a given analyte, was calculated for at least 2 treatment periods (where 1 of the treatment periods was the period in which the participant received the reference product [Treatment C]) and who had no major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
h*ng/mL
  Ticagrelor | 3462 (43.8) | 3423 (41.4) | 3546 (45.0)
  AR-C124910XX | 1488 (23.5) | 1441 (24.5) | 1513 (22.7)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Geometric Mean Ratio = 97.76, 90% CI 2-sided [94.46 to 101.18]
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Geometric Mean ratio = 96.38, 90% CI 2-sided [93.24 to 99.63]
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Statistical assessment of metabolite AR-C124910XX relative bioavailability following ticagrelor OD tablets administered compared to ticagrelor IR tablets; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 98.43, 90% CI 2-sided [94.75 to 102.25]
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 95.15, 90% CI 2-sided [91.59 to 98.85]

3. Primary Outcome: Area Under Plasma Concentration-time Curve From Zero to Infinity (AUC) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: Comparison of AUC (Area under plasma concentration-time curve from zero to infinity) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
ng*hr/mL
  Ticagrelor | 3520 (45.1) | 3485 (42.8) | 3606 (46.3)
  AR-C124910XX | 1547 (23.3) | 1503 (24.0) | 1573 (22.3)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Geometric Mean Ratio = 97.75, 90% CI 2-sided [94.40 to 101.21]
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 96.50, 90% CI 2-sided [93.31 to 99.80]
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 98.46, 90% CI 2-sided [94.85 to 102.20]
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 95.47, 90% CI 2-sided [91.99 to 99.08]

4. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: Comparison of tmax (Time to reach maximum observed concentration) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
hours
  Ticagrelor | 3.00 [1.00 to 4.02] | 3.00 [1.02 to 5.97] | 2.00 [1.00 to 6.00]
  AR-C124910XX | 3.07 [2.00 to 6.00] | 3.00 [2.00 to 6.02] | 3.00 [1.00 to 8.00]

5. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: Comparison of t½λz (half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
hours
  Ticagrelor | 7.74 (1.19) | 7.94 (1.19) | 7.86 (1.09)
  AR-C124910XX | 9.13 (1.91) | 9.12 (1.81) | 9.05 (1.68)

6. Secondary Outcome: Terminal Elimination Rate Constant (λz) of Ticagrelor and Its Active Metabolite, AR-C124910XX.
Description: Comparison of terminal elimination rate constant (λz) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
1/hour
  Ticagrelor | 0.0912 (0.0116) | 0.0889 (0.0116) | 0.0896 (0.0112)
  AR-C124910XX | 0.0792 (0.0170) | 0.0789 (0.0149) | 0.0794 (0.0160)

7. Secondary Outcome: Mean Residence Time (MRT) of Ticagrelor and Its Active Metabolite AR-C124910XX
Description: Comparison of MRT (mean residence time) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
hours
  Ticagrelor | 9.66 (2.14) | 10.1 (2.32) | 9.68 (2.47)
  AR-C124910XX | 13.3 (2.75) | 13.6 (2.90) | 13.2 (3.03)

8. Secondary Outcome: MRCmax (Ratio of Metabolite Cmax to Parent Cmax, Adjusted for Differences in Molecular Weights) of Active Metabolite AR-C124910XX
Description: Assessment of MRCmax (ratio of metabolite Cmax to parent Cmax, adjusted for differences in molecular weights) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
ratio | 0.340 (41.4) | 0.322 (44.8) | 0.327 (43.2)

9. Secondary Outcome: Ratio of Metabolite AUC(0-t) to Parent AUC(0-t), Adjusted for Differences in Molecular Weights (MRAUC [0-t]) of Active Metabolite AR-C124910XX
Description: Assessment of MRAUC(0-t) (Ratio of metabolite AUC(0-t) to parent AUC(0-t), adjusted for differences in molecular weights) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
ratio | 0.469 (42.3) | 0.460 (43.1) | 0.466 (44.0)

10. Secondary Outcome: Ratio of Metabolite AUC to Parent AUC, Adjusted for Differences in Molecular Weights (MRAUC) of Active Metabolite AR-C124910XX
Description: Assessment of MRAUC (Ratio of metabolite AUC to parent AUC, adjusted for differences in molecular weights) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
ratio | 0.480 (41.8) | 0.471 (42.9) | 0.476 (43.6)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. The term AE is used generally to include any AE whether serious or non-serious. A serious AE (SAE) is an AE that fulfills one or more of the following criteria: results in death, is immediately life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; is a congenital abnormality or birth defect; is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above.
Time Frame: From the date of randomization (Day 1 of the first treatment period) until the final follow-up visit (5 to 10 days after last administration of IMP).
Population: The safety analysis set included all participants who received at least 1 dose of ticagrelor and for whom any safety post-dose data were available.
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
Participants
  Participants with any AE | 3 | 4 | 3
  Participants with SAEs | 0 | 0 | 0

12. Secondary Outcome: Elimination Rate Constant (Kel) of Ticagrelor and Its Active Metabolite AR-C124910XX
Description: Comparison of kel (elimination rate constant) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet - when administered with and without water - and ticagrelor IR tablet. Blood samples for the determination of plasma concentrations of both ticagrelor and its active metabolite AR-C124910XX will be collected for each treatment period: 0 hours (pre-dose) and post-dose at 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
1/hour
  Ticagrelor | 0.0904 (1.15) | 0.0881 (1.15) | 0.0889 (1.14)
  AR-C124910XX | 0.0775 (1.23) | 0.0775 (1.21) | 0.0779 (1.21)

13. Secondary Outcome: Mean Change From Baseline for Vital Signs of Supine Blood Pressure (SBP) and Diastolic BP (DBP)
Description: The following variables were collected after the participants had rested in the supine position for at least 5 minutes: SBP and DBP.
Time Frame: Day 1 (pre dose, 2 hours, and 4 hours post dose) and Day 2 (24 hours post dose).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
mmHg
  SBP: Day 1, 2 hours post dose | 0 (8) | 0 (7) | 0 (8)
  SBP: Day 1, 4 hours post dose | 3 (8) | 0 (8) | 3 (7)
  SBP: Day 2, 24 hours post dose | 2 (8) | 1 (7) | 1 (8)
  DBP: Day 1, 2 hours post dose | -3 (5) | -2 (6) | -2 (6)
  DBP: Day 1, 4 hours post dose | -1 (6) | 0 (5) | -1 (6)
  DBP: Day 2, 24 hours post dose | 1 (6) | 1 (6) | -2 (6)

14. Secondary Outcome: Mean Change From Baseline for Vital Signs in Supine Pulse Rate.
Description: Vital signs i.e. Pulse (beats per minute [bpm]) were collected after the participant has rested in the supine position for at least 5 minutes.
Time Frame: At Screening and at Follow-up (these two examinations are 7 to 8 weeks apart) and during treatment periods at pre-dose and post-dose at 2, 4 and 24 hours.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
bpm
  Day 1, 2 hours post dose | 1 (5) | 3 (7) | 1 (4)
  Day 1, 4 hours post dose | 2 (6) | 4 (6) | 4 (6)
  Day 2, 24 hours post dose | 1 (5) | 2 (5) | 1 (4)

15. Secondary Outcome: Participants With Significant Findings in 12-Lead Electrocardiography (ECG).
Description: A 12-lead ECG was obtained after the participant rested in supine position for at least 10 minutes. The study physician was to judge the overall interpretation as normal or abnormal. If abnormal, it was decided as to whether or not the abnormality was clinically significant and the reason for the abnormality was recorded.
Time Frame: At Screening and at Follow-up (these two examinations are 7 to 8 weeks apart).
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
participants | 0 | 0 | 0

16. Secondary Outcome: Participants With Clinically Significant Findings in Hematology, Clinical Chemistry and Urinalysis.
Description: Participants were assessed through each laboratory variables for any significant abnormalities. Hematology assessments included white blood cell count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin and others. Clinical chemistry assessment included testing levels of sodium, potassium, urea, creatinine, albumin, calcium, glucose (fasting) and others. Urinalysis assessment included glucose, protein, blood and microscopy (if positive for blood or protein).
Time Frame: At Screening and at Follow-up (these two examinations are 7 to 8 weeks apart).
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 41 | 41 | 41
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of signing of informed consent (Day -28) up to 5-10 days after last administration of IMP (approximately 7-8 weeks).
Arm/Group | Treatment A | Treatment B | Treatment C
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 3/41 | 4/41 | 3/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=41) | Treatment B (N=41) | Treatment C (N=41)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.